CLINICAL TRIAL: NCT06075238
Title: Blinatumomab Prevents the Recurrence of Relapsed or Refractory Acute Lymphoblastic Leukemia After Allogeneic Hematopoietic Stem-cell Transplantation: A Prospective, Singlecentered, Single-arm, Phase II Clinical Study
Brief Title: Blinatumomab Prevents Recurrence of R/R ALL After Allo-HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-Blin 1.0
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Leukemia, Lymphoid
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blinatumomab (Experimental): Participants will take intravenous blinatumomab after allo-HSCT. The dose of one course was as follows: day 1-2: 8ug/day, continuous intravenous drip for 24 hours, day 3-7: 16ug/day, continuous intravenous drip for 24 hours. Treatment with blinatumomab was initiated within 60 to 90 days after transplantation and was administered bimonthly until 1 year after transplantation. Dexamethasone 20mg was administered 1 hour before administration on days 1 and 3 to prevent adverse events.
  Interventions: Drug: blinatumomab

INTERVENTIONS:
Drug: blinatumomab — The dose of one course was as follows: day 1-2: 8ug/day, continuous intravenous drip for 24 hours, day 3-7: 16ug/day, continuous intravenous drip for 24 hours. Dexamethasone 20mg was administered 1 hour before administration on days 1 and 3 to prevent adverse events.

SUMMARY:
The goal of this phase I/II clinical trial is to test in relapsed or refractory acute lymphoblastic leukemia (R/R ALL) patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer is:

• The efficacy and safety of blinatumomab maintenance therapy in reducing the recurrence rate a in R/R ALL patients after allo-HSCT. Participants will take intravenous blinatumomab after allo-HSCT. The dose of one course was as follows: day 1-2: 8ug/day, continuous intravenous drip for 24 hours, day 3-7: 16ug/day, continuous intravenous drip for 24 hours. Treatment with blinatumomab was initiated within 60 to 90 days after transplantation and was administered bimonthly until 1 year after transplantation. Dexamethasone 20mg was administered 1 hour before administration on days 1 and 3 to prevent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. B-ALL patients with history of relapse, or MRD positive in the last bone marrow examination before allo-HSCT;
2. Age ≥16 years old and ≤ 65 years old when signing informed consent Form (ICF);
3. KPS > 60 or ECOG 0-2;
4. The expected survival time is more than 3 months;
5. Complete remission (CR) after allo-HSCT with either myeloablative or non-myeloablative conditioning regimen determined by the investigator;
6. Reach the standard of hematopoietic reconstitution (neutrophil count

   ≥ 0.5×10^9/L for 3 consecutive days without G-CSF application, platelet count ≥ 20×10^9/L for 7 consecutive days without platelet transfusion, Hb ≥ 80 g /L without red blood cell transfusion); and neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 50×10^9/L within 45 days after transplantation;
7. No central nervous system involvement or clinical symptoms after transplantation;
8. Those who have no serious functional damage to important organs of the body;
9. Fully understand and be informed of this study and sign the ICF; willing to follow and have the ability to complete all test procedures;
10. Females of childbearing age must afford a serum pregnancy test within 7 days before the first dose, and the result should be negative; female participants and their partners should agree to use effective contraception from signing the ICF until 6 months after the last dose.

Exclusion Criteria:

1. Serious basic diseases of important organs: such as myocardial infarction, chronic cardiac insufficiency, decompensated hepatic insufficiency, renal function, gastrointestinal insufficiency, etc.;
2. Uncontrolled active infection (including bacterial, fungal, or viral infection), and drug treatment is ineffective;
3. Participating in other clinical studies, or planning to start treatment in this study and less than 4 weeks before the end of treatment in the previous clinical study;
4. Poor graft function (PGF) occurred after allo-HSCT;
5. Combined with other malignant tumors and require treatment;
6. Active GVHD;
7. Have a history of allergy to Chidamide;
8. Pregnant or lactating females;
9. Patients with known history of human immunodeficiency virus (HIV) virus infection and/or acquired immunodeficiency syndrome;
10. Patients with active chronic hepatitis B or active hepatitis C;
11. History of prolonged QT syndrome;
12. Patients considered by other researchers to be unsuitable for this study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival of this group of patients at the end of 2 year
100 day adverse events (AE) | Day +100
  non-hematologic adverse events

SECONDARY OUTCOMES:
Non-relapse mortality (NRM) | 6 months
  Non-relapse mortality of this group of patients at the end of 6 month
Relapse rate | 2 years
  Relapse rate of this group of patients at the end of 2 year
Overall survival (OS) | 2 years
  Overall survival of this group of patients at the end of 2 year
Cumulative incidence of acute graft versus host disease (aGVHD) | Day +100
  Cumulative incidence of acute graft versus host disease (aGVHD) of this group of patients at day+100
Cumulative incidence of chronic graft versus host disease (cGVHD) | 2 years
  Cumulative incidence of chronic graft versus host disease (cGVHD) of this group of patients at the end of 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No